CLINICAL TRIAL: NCT01795534
Title: Beetroot Juice as a Potential Ergogenic Aid During Exercise in Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Jan 13
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2015-03

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beetroot shot then placebo shot (Experimental): Intervention: Participants will first consume a Beetroot shot: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate) (Beet It, James White Drinks Ltd, Ipswich, UK).
  Following a four day wash out, participants will then consume a Nitrate-depleted beetroot shot: 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate)(Beet It, James White Drinks Ltd, Ipswich, UK)
  Interventions: Dietary Supplement: Beetroot shot then placebo shot
- Placebo shot then beetroot shot (Placebo Comparator): Intervention: Participants will first consume a Nitrate-depleted beetroot shot: 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate)(Beet It, James White Drinks Ltd, Ipswich, UK).
  Following a four day wash out, participants will then consume a Beetroot shot: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate) (Beet It, James White Drinks Ltd, Ipswich, UK).
  Interventions: Dietary Supplement: Placebo shot then beetroot shot

INTERVENTIONS:
Dietary Supplement: Beetroot shot then placebo shot — Beetroot shot, four day wash out, then placebo shot
  Arms: Beetroot shot then placebo shot
Dietary Supplement: Placebo shot then beetroot shot — Placebo shot, four day wash out, then beetroot shot
  Arms: Placebo shot then beetroot shot

SUMMARY:
The study will aim to describe and evaluate the effect of beetroot juice supplementation upon whole body running exercise at altitude. It is hypothesised that beetroot supplementation will decrease time to complete a 10 km time trial.

ELIGIBILITY:
Inclusion Criteria:

- Trained athletes with personal best performances for a 10km run of sub 40 minutes

Exclusion Criteria:

- Unable to give informed consent Unstable medical condition.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie H Macdonald, PhD, Principal Investigator — Bangor University
Locations (1):
- Bangor University, Bangor, Gwynedd, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Shot Then Beetroot Shot: Intervention: participants will first consume a Nitrate-depleted beetroot shot: 1x70ml nitrate-depleted beetroot Placebo shot (~0.003mmol of nitrate)(Beet It, James White Drinks Ltd, Ipswich, UK)
  Following a four day wash out, participants will then consume a Beetroot shot: 1x70ml concentrated NO-3 shot of rich Beetroot juice (~7mmol nitrate) (Beet It, James White Drinks Ltd, Ipswich, UK).
Period: First Intervention (First Shot)
Arm/Group | Beetroot Shot Then Placebo Shot | Placebo Shot Then Beetroot Shot
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Wash Out Period (4 Days)
Arm/Group | Beetroot Shot Then Placebo Shot | Placebo Shot Then Beetroot Shot
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (Second Shot)
Arm/Group | Beetroot Shot Then Placebo Shot | Placebo Shot Then Beetroot Shot
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes groups randomized to receive beetroot shot first and placebo first.
Groups:
- All Participants: Includes groups randomized to receive beetroot shot first and placebo first.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete a 10 km Run
Description: Time taken following consumption of beetroot shot or consumption of placebo shot
Time Frame: Period 1 (on day of 1st intervention) and period 2 (on day of 2nd intervention)
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Beetroot Shot: Includes groups randomized to receive beetroot first and placebo first.
  Data is for all participants following consumption of 1x70ml concentrated NO-3 shot of rich beetroot juice (~7mmol nitrate) (Beet It, James White Drinks Ltd, Ipswich, UK).
- Placebo Shot: Includes groups randomized to receive beetroot first and placebo first.
  Data is for all participants following consumption of 1x70ml nitrate-depleted beetroot shot (~0.003mmol of nitrate)(Beet It, James White Drinks Ltd, Ipswich, UK).
Arm/Group | Beetroot Shot | Placebo Shot
Number analyzed (Participants) | 10 | 10
Seconds | 2862 (233) | 2874 (265)

ADVERSE EVENTS:
Time Frame: During three study periods only (1st intervention, wash out period, second intervention)
Groups:
- Beetroot Shot: Data is for all participants following consumption of 1x70ml concentrated NO-3 shot of rich beetroot juice (~7mmol nitrate) (Beet It, James White Drinks Ltd, Ipswich, UK).
- Placebo Shot: Data is for all participants following consumption of 1x70ml nitrate-depleted beetroot shot (~0.003mmol of nitrate)(Beet It, James White Drinks Ltd, Ipswich, UK).
Arm/Group | Beetroot Shot | Placebo Shot
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes